CLINICAL TRIAL: NCT03008902
Title: A Cross-sectional Study Using Motion Analysis to Determine Whether Age and Hyperkyphosis Are Associated With Thoracic Spine Motion and Loading
Brief Title: A Study of Effects of Age and Hyperkyphosis on Spine Motion and Loading
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: University of Denver (Other)
Responsible Party: Principal Investigator, Dennis Anderson, Staff Scientist II, Beth Israel Deaconess Medical Center
Other Study IDs: 2015P000394
Record Dates: First submitted 2016-12-16; First posted 2017-01-04 (Estimated); Last update posted 2018-10-04 (Actual); Status verified 2018-10

CONDITIONS: Kyphosis; Vertebral Fracture
MeSH Terms: conditions — Kyphosis; Spinal Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-patients: Non-patients, who have not had vertebral fractures or hyperkyphosis, and have not been seen at BIDMC, will be recruited from the community as described in section B3C and B6 below. The non-patient group will consist of 16 healthy adults ages 18-40.
  Interventions: Procedure: Near-infrared passive motion capture recording
- Patients: Patients, who have been seen at BIDMC for vertebral fractures or hyperkyphosis, will be identified by review of medical records as described in B3C and B6 below. The patient group will consist of 32 adults ages 75 and older who have previously been diagnosed with a thoracic vertebral fracture at BIDMC.
  Interventions: Procedure: Near-infrared passive motion capture recording

INTERVENTIONS:
Procedure: Near-infrared passive motion capture recording — Full body movement will be recorded during movements using near infrared passive motion capture. This procedure is non-invasive and standard practice in biomechanics labs. Movement will be recorded using an eight-camera system. Retroreflective markers are placed at strategic joint locations to characterize limb movement. Accuracies of the marker positions are sub-millimeter, and allow accurate characterization of limb rotation and translation during movements. Passive reflective marker clusters (3 markers each) will be attached to subjects at 8 locations along the spine. Additional markers will be applied to the manubrium of the sternum, head, pelvis, and extremities. Eight EMG surface electrode pairs will be used to record activation from the left and right erector spinae, latissimus dorsi, trapezius and rectus abdominis muscles during all motions.

SUMMARY:
We are studying how spine movement changes with age, and when people have vertebral fractures (cracks in the bones of the spine) or hyperkyphosis (a forward stooped posture).

DETAILED DESCRIPTION:
The purpose of this study is to obtain unique measures of thoracic spinal motion in young, older, and hyperkyphotic older adults. We will then develop unique subject-specific musculoskeletal models of these individuals to estimate loads applied to the vertebrae in vivo, and examine how spinal motion and loading vary with age and increased kyphosis.

Vertebral fractures (VFs) are the most common type of fracture in older adults, occurring in 20-35% of women and 15-25% of men over the age of 50, and are associated with significant morbidity, increased mortality, and annual costs exceeding $1 billion in the United States. However, limited understanding of the mechanisms (beyond low vertebral bone mineral density and strength) that lead to VFs hinders our ability to predict and prevent these injuries.

Similarly, hyperkyphosis, defined as excess forward curvature of the thoracic spine, is suffered by 20-40% of older adults, but its causes are poorly understood and it has no standard clinical treatment. Hyperkyphosis and VFs are inter-related, as individuals with VFs often have worse kyphosis, while hyperkyphosis is an independent risk factor for future VFs. Hyperkyphosis may increase VF risk through increased vertebral loading, but better understanding is needed of the biomechanics of this common spine condition.

VFs occur more often at mid-thoracic (T7-T8) and thoraco-lumbar (T12-L1) vertebrae than elsewhere in the spine, and it has been suggested that biomechanical factors predispose these areas to fracture by increasing vertebral loading. In the first phase of this project, a novel musculoskeletal model was developed that uniquely predicts peaks in vertebral loading around the T12-L1 region of the spine, but this was not observed in the mid-thoracic region. Our preliminary data suggested that increased thoracic stiffness causes greater vertebral loading at mid-thoracic levels (T7-T9), while increased thoracic kyphosis increases vertebral loading, particularly in the thoraco-lumbar (T12-L1) region.

Further advances in musculoskeletal modeling will are needed to fully evaluate these possibilities, but a particular knowledge gap remains regarding the in vivo kinematics of the thoracic spine and ribcage in both healthy and hyperkyphotic individuals. This project aims to fill that gap by producing novel in vivo measurements of thoracic spine motion in young, older, and hyperkyphotic older adults.

ELIGIBILITY:
No exclusion criteria shall be based on race, ethnicity, or sex.

Inclusion Criteria (Non-patient group):

* Males and females, ages 18 - 40 years
* Able to perform activities such as walking, standing, sitting, bending or lifting without assistance
* Willing to sign informed consent form

Exclusion Criteria (Non-patient group):

• Conditions that might alter thoracic biomechanics: Examples of these include scoliosis, a history of traumatic thoracic injury or spinal surgery, neuromuscular conditions such as Parkinson's disease or muscular dystrophy.

* Body mass index > 30 kg/m2
* Pregnancy
* Latex allergies
* Currently taking muscle relaxers, steroids, or narcotics
* Participation in another research study with radiation exposure
* Previous exposure to radiation as part of a medical procedure in the past six months
* Musculoskeletal injury or condition that is currently affecting normal activity or movement. Examples of this could include sprains, strains, dislocations or fractures that prevent one from walking, standing, sitting, bending or lifting in a normal manner.

Inclusion Criteria (Patient group):

* Males and females, ages 75 years and older.
* Patients who received a lateral thoracic spine x-ray and had a diagnosis of a vertebral fracture (ICD9 - 805.2) in the year 2011 or later.
* At least 6 months since diagnosis of vertebral fracture.
* Measurable T4-T12 Cobb angle in lateral thoracic spine x-ray.
* Currently living in the Boston area.
* Able to perform activities such as walking, standing, sitting, bending or lifting without assistance
* Willing to sign informed consent form

Exclusion Criteria (Patient group):

• Conditions (unrelated to vertebral fracture and hyperkyphosis) that might alter thoracic biomechanics: Examples of these include scoliosis, a history of traumatic thoracic injury or spinal surgery, neuromuscular conditions such as Parkinson's disease or muscular dystrophy.

* Body mass index > 30 kg/m2
* Latex allergies
* Currently taking muscle relaxers, steroids, or narcotics
* Musculoskeletal injury or condition that is currently affecting normal activity or movement. Examples of this could include sprains, strains, dislocations or fractures that prevent one from walking, standing, sitting, bending or lifting in a normal manner.
* A score ≥10 on the Short Blessed Test, suggesting possible impaired cognitive function or dementia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Non-patients
  Non-patients, who have not have not been seen at BIDMC for vertebral fractures or hyperkyphosis, will be recruited from the local community. The non-patient group will consist of 16 healthy adults ages 18-40.
  Patients
  Patients, who have been seen at BIDMC for vertebral fractures or hyperkyphosis, will be identified by review of medical records. The patient group will consist of 32 adults ages 75 and older who have previously been diagnosed with a thoracic vertebral fracture at BIDMC.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2017-04-18 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Thoracic spine range of motion, in degrees. | Day 1
  Full body movement will be recorded during subject movements using near infrared passive motion capture. This procedure is non-invasive and standard practice in biomechanics labs. Passive reflective marker clusters will be attached to subjects along the spine at T1, T4, T5, T8, T9, T12, L1, and additional markers will be applied to the manubrium of the sternum, head, pelvis, and extremities. Marker positions during subject movements will be recorded with sub-millimeter accuracy using an eight-camera system from Vicon Motion Systems (Centennial, CO). Recorded marker positions will be applied to a musculoskeletal model of the subject through an inverse kinematics algorithm in order to provide estimates of thoracic spine angular range of motion in flexion-extension, lateral bending, and axial rotation during each subject movement.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Anderson, Ph.D., Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No